CLINICAL TRIAL: NCT05925894
Title: Efficacy of the Intracamerally Administered Mydriatics for Cataract Surgery in Patients With Primary Open-angle Glaucoma.
Brief Title: Efficacy Mydrane ® for Cataract Surgery in Patients With Concomitant Primary Open Angle Glaucoma.
Acronym: MIGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Ricci Francesco, Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4654
Record Dates: First submitted 2023-02-01; First posted 2023-06-29 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Cataract Surgery
Keywords: mydriasis and intraocular anaesthesia
MeSH Terms: conditions — Mydriasis | interventions — Anesthetics

STUDY DESIGN:
Intervention Model Description: In this retrospective study, we collected pre- and post-operative data from 60 patients who underwent elective cataract extractions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Mydriatic Eyedrops (Active Comparator): Group 1 patients included instillation of one drop each of tropicamide 0.5% and phenylephrine 10% ( VISUMIDRIATIC FENILEFRINA) at 30, 20, and 10 min prior to surgery.
  Interventions: Drug: Efficacy of a Standardized Intracameral Combination of Mydriatics and Anesthetic (Mydrane ®) for Cataract Surgery in Patients With Concomitant Primary Open Angle Glaucoma
- Group 2: Insert Device Mydriasert® (Experimental): Group 2 patients had the Mydriasert® (Phenylephrine Hydrochloride,Tropicamide) device placed in the inferior conjunctival sac at least 1 h before surgery
  Interventions: Drug: Efficacy of a Standardized Intracameral Combination of Mydriatics and Anesthetic (Mydrane ®) for Cataract Surgery in Patients With Concomitant Primary Open Angle Glaucoma
- Group 3: Intracameral Anesthesia Mydrane® (Experimental): Group 3 patients received 0.2 mL intracameral Mydrane®(0.2 mg/ml + 3.1 mg/ml + 10 mg/ml tropicamide, lidocaine hydrochloride, phenylephrine hydrochloride) immediately following the clear corneal incision; the surgeon allowed 45-60 s for adequate pupil dilation before performing continuous curvilinear capsulorhexis (CCC)
  Interventions: Drug: Efficacy of a Standardized Intracameral Combination of Mydriatics and Anesthetic (Mydrane ®) for Cataract Surgery in Patients With Concomitant Primary Open Angle Glaucoma

INTERVENTIONS:
Drug: Efficacy of a Standardized Intracameral Combination of Mydriatics and Anesthetic (Mydrane ®) for Cataract Surgery in Patients With Concomitant Primary Open Angle Glaucoma — 60 patients with coexisting POAG and cataract who underwent elective cataract extraction. All patients underwent ophthalmic routine examinations including automatic visual field examination, anterior chamber configuration, specular microscopy and arterial blood pressure measurement prior to surgery, 24 hours and 30 days postoperatively. All cataract surgeries were videorecorded, and all measurements were performed using media player. 20 patients received topical mydriatic eye drops, 20 patients received Mydriasert ® whereas 20 patients received intracameral injection of Mydrane ® just after the first incision.

SUMMARY:
The aim of this study is to compare Mydrane ®, mydriatic eye drops and Mydriasert ® in terms of pupil site stability, surgical time, visual field and anterior chamber configuration modifications among primary open angle glaucoma (POAG) patients during cataract extraction surgery.

DETAILED DESCRIPTION:
60 patients with coexisting POAG and cataract who underwent elective cataract extraction. All patients underwent ophthalmic routine examinations including automatic visual field examination, anterior chamber configuration, specular microscopy and arterial blood pressure measurement prior to surgery, 24 hours and 30 days postoperatively. All cataract surgeries were videorecorded, and all measurements were performed using media player. 20 patients received topical mydriatic eye drops, 20 patients received Mydriasert ® whereas 20 patients received intracameral injection of Mydrane ® just after the first incision.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years of age
* diagnosed with age-related cataract with concomitant POAG well controlled by pharmacological therapy (IOP within its target during the entire day in a minimum of 12-month follow-up with constant use of anti-glaucoma medications)
* required cataract extraction under local anesthesia
* no history of previous surgery in the study eye

Exclusion Criteria:

* patients with POAG requiring glaucoma surgery
* ocular trauma or infection
* other forms of glaucoma
* pseudo-exfoliation and exfoliation syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-12-18 (Actual); Study Completion 2022-01-09 (Actual)

PRIMARY OUTCOMES:
Stability of mydriasis | 1 hour
  All cataract surgeries were video-recorded, and all measurements were performed using media player software (VideoLAN Non-Profit Organization, Paris, France) with two different operators (M.R. and F.R.) based on the images acquired immediately prior to the corneal incision (T1), injection of the ophthalmic viscosurgical device (OVD) (T2), capsulorhexis (T3), IOL insertion (T4), and cefuroxime injection (end of surgery) (T5). The pupil size immediately prior to the capsulorhexis was defined as the maximum mydriasis. We recorded all the surgery with OPMI LUMERA® 700 ZEISS and then measured with media player software all the pupil size.
Duration of surgery | 1 hour
  mean duration of surgery, All cataract surgeries were video-recorded, and all measurements were performed using media player software (VideoLAN Non-Profit Organization, Paris, France) with two different operators (M.R. and F.R.) based on the images acquired immediately prior to the corneal incision (T1), injection of the ophthalmic viscosurgical device (OVD) (T2), capsulorhexis (T3), IOL insertion (T4), and cefuroxime injection (end of surgery) (T5).

SECONDARY OUTCOMES:
Pain experience | up to 4 weeks
  Patients were asked to complete a questionnaire using the the Visual Analogue Scale (VAS) scale to evaluate surgical pain related to the procedure. The scale simply consists of a 10 cm strip of paper which has two "end points" at the ends which are defined as "no pain" and "the worst pain I can imagine".
Central corneal thickness (CCT) and corneal endothelium cell density (CD) changes | up to 4 weeks
  Specular microscopy values were evaluated by using the Perseus (CSO, Italy) The Perseus specular microscope is a non-contact automated instrument with auto alignment and a touch screen that automatically conducts studies for measuring endothelial cell layer density using the corner method to analyze the endothelial cells. The instrument has a reliability index that evaluates the quality of acquisition, this is based on a calculation of the percentage of the total endothelium area relative to the maximum number of countable endothelial cells per field (edited area). Corneal endothelial cell density (CD) is calculable using a units of measure based on cells/mm2.
Visual field defects | up to 4 weeks
  The 30-2 SITA STANDARD algorithm (HFAII740: Humphrey Field Analyzer II; Carl Zeiss Meditec, Dublin, California, USA) was used for the standard automatic visual field examination of all the patients to investigate the visual field defects, mean deviation (MD), and pattern standard deviation (PSD) modifications at baseline and 30 days postoperatively. Visual field testing was performed with visual correction in a dark room.
Anterior segment parameters variations | up to 4 weeks
  Anterior chamber depth (ACD) and both nasal and temporal iridocorneal angles were measured by a single experienced operator who obtained a horizontal scan, including sections of the nasal and temporal quadrants of all the patients, using AS-OCT (Visante, software version 2.01.88; Carl Zeiss Meditec, Dublin, CA) in a dark room with the images centered on the pupil . High-resolution images were taken in the anterior segment single-scan mode along the horizontal meridian with the subjects seated.When the corneal reflex was visible, the image was captured. ACD (from the corneal endothelium to the anterior surface of the crystalline lens) were then measured (ACD was obtained using the on-screen calibrated caliper function).

CONTACTS AND LOCATIONS:
Overall Officials: francesco ricci, Principal Investigator — Policlinico Gemelli
Locations (1):
- Policlinico Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Labetoulle M, Behndig A, Tassignon MJ, Nuijts R, Mencucci R, Guell JL, Pleyer U, Szaflik J, Rosen P, Berard A, Chiambaretta F, Cochener-Lamard B; Intracameral Mydrane (ICMA), Ethics Group. Safety and efficacy of a standardized intracameral combination of mydriatics and anesthetic for cataract surgery in type-2 diabetic patients. BMC Ophthalmol. 2020 Mar 3;20(1):81. doi: 10.1186/s12886-020-01343-x. PMID 32126990